CLINICAL TRIAL: NCT03966820
Title: Subjective Ageing in Fibromyalgia: Why Fibromyalgia Patients Feel Old?
Brief Title: Subjective Ageing in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH3
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
Keywords: Anxiety; Cognitive ageing; Depression; Fatigue; Fibromyalgia; Quality of life; Sleep
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjective age or felt age is the term used for how the person feels; one can feel same, younger or older than their actual age. Feeling younger or feeling older may be associated with depression, anxiety, fatigue, sleep, quality of life or cognitive function.

DETAILED DESCRIPTION:
In this cross-sectional study, the investigators hypothesized that fibromyalgia patients mostly feel older than their actual age and this felt age may be associated with depression, anxiety, fatigue, sleep, quality of life or cognition. After power analysis, study sample calculated as 262 patients, the present study will use 2016 revised American College of Rheumatology criteria to diagnose fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis using 2016 revised American College of Rheumatology
* aged >18 years old
* Widespread pain more than 3 months

Exclusion Criteria:

* Any disease that can cause depression, anxiety, fatigue, poor sleep quality or poor cognitive function except from fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 262 patients diagnosed with fibromyalgia will be included in the study
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Subjective age | Four months
  The study will ask the patient: " how old do you feel?". Subjective age will calculate as Subjective age extracted from actual age. If the result is positive, the patient feel younger, if visa versa the patient feels older
Depression | Four months
  The status of depression will calculate using Beck Depression Inventory. This inventory is a self scored, 21 item questionnaire. Higher scores indicate higher depression levels of the patient.
Anxiety | Four months
  The status of anxiety will calculate using Beck Anxiety Inventory. This inventory is a self scored, 21 item questionnaire. Higher scores indicate higher anxiety levels of the patient. The total score is calculated by finding the sum of the 21 items. Each question scored 0 to 3 points. Score of 0-21 = low anxiety,score of 22-35 = moderate anxiety, score of 36 and above = potentially concerning levels of anxiety
Sleep | Four months
  The status of sleep quality of the patients will calculate using Pittsburgh Sleep Quality Index. The index is a self- scored 24 item questionnaire and 7 subgroups. Higher scores show bad sleep quality and lower scores indicate good sleep quailty.
Fatigue | Four months
  The fatigue levels of the patients will be determined using The Fatigue Severity Scale. This scale self-reported 9 item questionnaire, each question scored between 0-7, total score divided to nine and if the result <2.8, no fatigue and if > 6.1, chronic fatigue syndrome diagnosis can be made. Higher score shows higher probability of chronic fatigue syndrome.
Cognitive Function | Four months
  The cognition status of the patients will be determined using Mini-mental State Examination. This test includes five subscales, scoreing 0 - 30 points. Lower scores show poorer cognitive function
Life Quailty | Four months
  The quality of life of the patients will be determined using Short-form 36. The self-reported questionnaire includes 11 subscales. Higher scores show poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Guler, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No